CLINICAL TRIAL: NCT06084117
Title: High Flow Nasal Oxygen For Hypercapnic, Acidotic Exacerbation Chronic Obstructive Pulmonary Disease
Brief Title: High Flow Nasal Oxygen for Exacerbation COPD
Acronym: HiCAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Franciscus Gasthuis (Other)
Collaborators: Reinier de Graaf Groep (Other); Haga Medisch Centrum (Unknown); Ikazia Hospital, Rotterdam (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HiCAP
Record Dates: First submitted 2023-10-02; First posted 2023-10-16 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Acute Exacerbation of COPD

STUDY DESIGN:
Intervention Model Description: pilot randomized unblinded controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High Flow Nasal Oxygen (HFNO) (Experimental): Patients will start at a flow of 50 L/min and a temperature of 37°C, FiO2¬ will start at 25%, and titrated to target SpO2 (88-92%, as in usual care).
  Interventions: Other: HFNO
- Non-Invasive Ventilation (NIV) (Active Comparator): Patients will be started at
  * Using the facemask interface: EPAP/PEEP set at 5-7 cmH2O and PS of 5-7 cmH2O (equal to IPAP of 10-14 cmH2O).
  * Using the helmet interface; EPAP/PEEP set at least 10 cmH2O and PS of 10 cmH2O (equal to IPAP of 20 cmH2O).
  * PEEP/EPAP and IPAP/PS can be titrated to effectiveness, tolerance and comfort
  * FiO2 should be set to achieve a SpO2 of 88-92%
  Interventions: Other: NIV

INTERVENTIONS:
Other: HFNO — Respiratory support with HFNO (as opposed to NIV, as per standard of care)
  Arms: High Flow Nasal Oxygen (HFNO)
Other: NIV — Respiratory support with Non-invasive ventilation, standard of care
  Arms: Non-Invasive Ventilation (NIV)

SUMMARY:
In this pilot study the feasibility of performing a larger trial to study the non-inferiority of High Flow Nasal Oxygen compared to non-invasive ventilation in patients with acute acidotic hypercapnic exacerbation of COPD wil be investigated

DETAILED DESCRIPTION:
Rationale: Chronic Obstructive Pulmonary Disease (COPD) is frequently complicated by a worsening of symptoms, known as acute exacerbations (AECOPD). These exacerbations can result in a life-threatening condition with an impaired gas exchange, resulting in hypercapnia and as a result respiratory acidosis. The current standard of care of respiratory support for these patients is non-invasive ventilation (NIV), which has been shown to reduce morbidity and mortality. However, NIV is often unsuccessful, due to intolerance, agitation or patient-ventilation dyssynchrony. Furthermore, NIV is a resource-intensive therapy. High flow nasal oxygen (HFNO) is a non-invasive respiratory support mode that provides heated and humidified gas through soft nasal prongs. Several studies have shown that HFNO improves gas exchange and reduces work of breathing in non-hypercapnic respiratory failure. Furthermore, HFNO is thought to be better tolerated than NIV and the nursing effort may be lower compared to NIV. The hypothesis is that HFNO is non-inferior to NIV for patients with acidotic, hypercapnic AECOPD regarding the need for intubation and mortality, and that it increases patient comfort and reduces nursing effort.

Objective: To assess the feasibility of a larger study comparing HFNO with NIV as first line treatment in hypercapnic, acidotic AECOPD.

Study design: prospective, randomized, multi-center, unblinded, pilot study. Study population: Patients with acidotic, hypercapnic AECOPD Intervention (if applicable): HFNO versus NIV as first line treatment at presentation Main study parameters/endpoints: Feasibility: screening rate, inclusion rate, feasibility as qualified by staff and nurses.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: All participating patients will receive standard of care (i.e., admission to the monitored ward or ICU for intensive monitoring and regular blood withdrawals, steroids, bronchodilator inhalation therapy). There will be one extra questionnaire after 3 months, but no extra blood samples or site visits, compared to regular care for the participating patients. Permission of the patient will be obtained to register date of hospital discharge and outcome after ICU discharge and ask them to fill out questionnaires at 3 months after admission about their quality of life. Previous studies have not shown that HFNO is inferior to NIV with regards to outcomes (intubation rate, mortality), albeit that they were not powered to prove non-inferiority.

ELIGIBILITY:
Inclusion Criteria:

* Known chronic obstructive pulmonary disease
* Acute hypercapnic exacerbation of this condition, defined as: PaCO2>45 mmHg or >6.0 kPa and pH 7.20-7.35
* Age >40 years

Exclusion Criteria:

* Asthma
* Immediate need for intubation, based on clinical judgement of the attending physician.
* Impossibility to apply either one of the two interventions
* Patient not expected to give immediate or delayed informed consent (e.g. known cognitive impairment, dementia, active serious psychiatric disease, mental retardation).
* Established home-NIV or home CPAP, known indication for home-NIV or CPAP (e.g. OSAS or obesitas hypoventilation syndrome).
* Impeding death
* Concurrent (respiratory) diseases that may influence treatment efficacy: acute heart infarction, cardiogenic lung edema, massive pulmonary embolism (intermediate-high risk or more). NB; pulmonary infections (viral and bacterial) are a common cause of exacerbation and are no reason for exclusion.
* Other acute diseases that preclude participation in the trial such as hemodynamic instability (need for vasopressors), reduced consciousness with need for intubation, severe intoxication
* Tracheostomized patients
* Participation in other interventional trials
* Impossibility to admit the patient to the participating ICU or monitored ward (e.g. medium care / high dependency unit, depending on local infrastructure).
* Previous explicit (or written) objection to participation in research - bicarbonate <20 mmol/L

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-14 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
feasilibity to perform a larger RCT inclusion rate | 1 year
  Inclusion rate
feasibility to perform a larger RCT screening rate | 1 year
  Screening rate
feasibility to perform a larger RCTperceived | 1 year
  perceived feasibility as qualified by staff and nurses
feasibility to perform a larger RCT protocol deviations | 1 year
  protocol deviations

SECONDARY OUTCOMES:
Treatment failure | 30 days
  cross-over, invasive mechanical ventilation, death
duration of intervention | 30 days
  time of respiratory support
need for sedation | untill end of ICU admission
  use of sedatives, and type of sedation
heart rate | at start, 1, 2, 6, 12, 24 and every 24 hours untill discharge
  beats per minute
respiratory rate | at start, 1, 2, 6, 12, 24 and every 24 hours untill discharge
  breaths per minute
blood pressure | at start, 1, 2, 6, 12, 24 and every 24 hours untill discharge
  systolic and diastolic pressure in mmHg
SpO2 | at start, 1, 2, 6, 12, 24 and every 24 hours untill discharge
  peripheral saturation by pulsoxymeter (in %)
blood gas | at start, 1, 2, 6, 12, 24 and every 24 hours untill discharge
  with pH, PO2, PCO2, bicarbonate
dyspnea score | at start, 1, 2, 6, 12, 24 and every 24 hours untill discharge
  Borg dyspnea score (0-10 on VAS)
Clinical Parameters | at start, 1, 2, 6, 12, 24 and every 24 hours untill discharge
  heart rate, respiratory rate, blood pressure, Spo2, arterial blood gas, dyspnea score, glasgow coma scale, RASS, seceretions
consciousness | at start, 1, 2, 6, 12, 24 and every 24 hours untill discharge
  glasgow coma scale (EMV)
agitation and sedation level | at start, 1, 2, 6, 12, 24 and every 24 hours untill discharge
  Richmond Agitation and Sedation scale (RASS)
secretions | at start, 1, 2, 6, 12, 24 and every 24 hours untill discharge
  (as 0 (absent), 1 (low quantity), 2 (intermediate), 3 (abundant), or 4 (very abundant) little to normal/abundant)
HFNO ventilatory support parameters flow | at start, 1, 2, 6, 12, 24 and every 24 hours untill discharge
  flow in L/min
HFNO ventilatory support parameters FiO2 | at start, 1, 2, 6, 12, 24 and every 24 hours untill discharge
  FiO2 in %
HFNO ventilatory support parameters temperature | at start, 1, 2, 6, 12, 24 and every 24 hours untill discharge
  temperature in Celcius
NIV ventilatory support parameters PEEP | at start, 1, 2, 6, 12, 24 and every 24 hours untill discharge
  PEEP in cmH2O
NIV ventilatory support parameters PS | at start, 1, 2, 6, 12, 24 and every 24 hours untill discharge
  PS in cmH2O
NIV ventilatory support parameters: FiO2 | at start, 1, 2, 6, 12, 24 and every 24 hours untill discharge
  FiO2 in %
(dys)comfort score | at start, 1, 2, 6, 12, 24 and every 24 hours untill discharge
  10 point VAS scale
HACOR score | at start, 1, 2, 6, 12, 24 and every 24 hours untill discharge
  calculated from abovementioned parameters (pH, conciousness, PaO2/Fio2, respiratory rate)
facial pressure sores | at start, 1, 2, 6, 12, 24 and every 24 hours untill discharge
  scored daily: yes or no, and if yes: grade 1-4
nursing effort | first 6 hours of study
  respiratory support interventions per 2 hour by peat list
nursing effort VAS | at start, 1, 2, 6, 12, 24 and every 24 hours untill discharge
  experienced nursing effort at a VAS scale from 1-10
30d mortality | 30 days
  mortality
90d mortality | 90 days
  mortality
90d quality of life EQ5D | 90 days
  EQ5D
90d quality of life SF36 | 90 days
  SF-36
90d anxiety and depression | 90 days
  HADS
90d PTDS | 90 days
  IES-R
90d PTSD | 90 days
  IES-R
90d dyspnea CCQ | 90 days
  CCQ
90d dyspnea MRC | 90 days
  MRC
need for intubation and mechanical ventilation | during ICU admission
  intubation
need for switch to other modality | during ICU admission
  cross over to NIV from HFNO or from HFNO to NIV
reason of treatment failure | during ICU admission
  reason of treatment failure: clinical deterioration, failure to improve, other.
expression of treatment failure | during ICU admission
  worsening of pH, PaCO2, respiratory rate, consiousness, agitation/discomfort, other

CONTACTS AND LOCATIONS:
Overall Officials: Dorien Kiers, MD, PhD, Principal Investigator — Franciscus Gasthuis & Vlietland
Locations (4):
- Netherlands (4):
  - Reinier de Graaf, Delft
  - Franciscus Gasthuis & Vlietland, Rotterdam
  - Ikazia, Rotterdam
  - Haaglanden Medisch Centrum, The Hague

IPD SHARING:
Plan to Share IPD: No